CLINICAL TRIAL: NCT07339319
Title: Treatment and Outcome of Patients With Mild Head Injury: a Retrospective Multicentre Study in Emilia Romagna
Brief Title: Treatment and Outcome of Patients With Mild Head Injury
Acronym: BTER23
Status: Recruiting | Type: Observational
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Other Study IDs: 1/2024/OSS/AUSLRE
Record Dates: First submitted 2026-01-05; First posted 2026-01-14 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Head Injury Trauma
Keywords: isolated head injury; First Aid; brain CT scan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
The study aims to assess the incidence of complications, such as intracranial haemorrhages and neurological deficits, in patients with head trauma treated in the emergency departments of the Emilia-Romagna Region and to compare the prognostic accuracy of the Canadian CT Head Rule and NEXUS Head CT Instrument in predicting post-traumatic complications. This is a retrospective multicentre cohort study that includes patients aged 18 years or older with isolated head trauma who underwent brain CT within 24 hours of the trauma. The data, sourced from hospital databases, will include medical history, prognostic scores, instrumental examinations, pharmacotherapy and adverse events. The primary objective is to determine the incidence of complications in patients who require surgery or who die, while the secondary objectives aim to compare the prognostic effectiveness of the two instruments in predicting complications. In addition, the study will examine the management strategies adopted and seek to identify any predictors of complications not included in current prognostic models. The results will contribute to improving the management of head trauma in emergency departments and optimising the use of available prognostic tools.

DETAILED DESCRIPTION:
Head trauma is one of the main causes of visits to the emergency room and hospitalisation. Globally, it is estimated that there are approximately 50 million cases of head trauma each year. In the United Kingdom, it is the leading cause of death and disability in patients under the age of 40. In Italy, according to SINCH data, approximately 250 patients per 100,000 inhabitants are hospitalised for head trauma each year, with a mortality rate of 17 cases per 100,000 inhabitants per year.

Although numerous guidelines have been drawn up for the management of patients with head trauma, the lack of high-quality studies limits the effectiveness of the recommendations, leading to heterogeneous management from a diagnostic and therapeutic point of view.

The main objective of this multicentre, retrospective cohort study is to assess the incidence of complications in patients with head trauma who attend the emergency departments of the Emilia-Romagna Region. The complications considered include intracranial haemorrhages of any nature and neurological deficits that may require surgery and/or lead to death. The study also aims to compare and validate the prognostic accuracy of the Canadian CT Head Rule and the NEXUS Head CT Instrument in predicting post-traumatic complications, as found by brain computed tomography (CT) performed in the emergency department.

Furthermore, the study compares the different management strategies adopted and assesses the presence of additional predictive factors for the onset of meta-traumatic complications, not covered by the prognostic tools used.

To achieve these objectives, the study plans to include adult patients (aged ≥18 years) capable of providing informed consent, who have been assessed in the Emergency Department with a diagnosis of isolated head trauma and subsequently discharged home or transferred to the OBI (Short-Term Intensive Care), Emergency Medicine, or other hospital wards. Patients must have undergone a brain CT scan during their diagnostic-therapeutic pathway and arrived at the Emergency Department within 24 hours of the trauma. The study will record data relating to medical history (recent and remote), pharmacological management (with particular attention to the use of antiplatelet or anticoagulant therapies), criteria for calculating the Canadian CT Head Rule score (a validated tool that helps to reliably rule out the presence of intracranial lesions requiring neurosurgical intervention without resorting to a CT scan) and the NEXUS Head CT Instrument (a tool used to predict the need for brain CT in patients with closed head injury). Vital signs, instrumental and laboratory tests, medications administered (with dosage and method of administration), and any adverse events will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18 years or older capable of self-determination
* patients assessed in the emergency department with a final diagnosis of isolated head trauma, subsequently discharged home or transferred to the OBI, Emergency Medicine and/or possibly admitted to other wards, who have undergone at least one brain CT scan during their diagnostic-therapeutic pathway
* GCS 13-15
* presentation <24 hours after trauma

Exclusion Criteria:

* patients aged < 18 years
* patients with multiple fractures outside the cranium
* patients with head trauma who have not undergone a brain CT scan
* GCS <13

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged ≥18 years, assessed in the Emergency Department with a diagnosis of isolated head trauma, who have undergone a brain CT scan within 24 hours of the trauma.
Sampling Method: Non-Probability Sample
Enrollment: 4500 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of complications following severe head trauma | 12 months
  To assess the incidence of complications, such as intracranial haemorrhages and neurological deficits, in patients with head trauma who require surgery and/or are at risk of death.

SECONDARY OUTCOMES:
Prognostic Accuracy of the Canadian CT Head Rule and the NEXUS Head CT Instrument in Predicting Post-Traumatic Complications | 12 months
  Evaluate the prognostic accuracy of the Canadian CT Head Rule and the NEXUS Head CT Instrument in predicting post-traumatic complications with Positive Predictive Value (PPV): Probability that patients identified as "high risk" will develop complications.
Comparison of management strategies in the Emergency Department | 12 months
  Compare the management strategies adopted in the Emergency Department for severe head trauma and identify predictive factors not considered by prognostic tools.

CONTACTS AND LOCATIONS:
Locations (4):
- Italy (4):
  - Ospedale Maggiore di Bologna, Bologna
  - Ospedale Sant'Orsola di Bologna, Bologna
  - Ospedale di Ferrara, Modena
  - AziendaUSL IRCCS Reggio Emilia, Reggio Emilia